CLINICAL TRIAL: NCT03932669
Title: Effect of Nilotinib in Cerebellar Ataxia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1811-074-985
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Ataxia, Cerebellar; Ataxia, Progressive
Keywords: spinocerebellar ataxia; treatment; nilotinib; bcr-abl; receptor-tyrosine-kinase-inhibitor
MeSH Terms: conditions — Cerebellar Ataxia; Ataxia; Spinocerebellar Ataxias | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib group (Experimental): Patients with SCA and taking nilotinib treatment
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 150-300mg daily dose of nilotinib

SUMMARY:
This is an institutional cohort study. Patients confirmed with spinocerebellar ataxia (SCA) and taking or planning to take Nilotinib (Tasigna®) are enrolled in this study. The daily dose of Nilotinib is 150mg-300mg and the patients will be followed up at 1, 3, 6, and 12 months. Rating scale for Friedreich's ataxia I and II and Barthel index are used as general function and daily living performance index. Scale for assessment and rating of ataxia (SARA) are used as an objective measure of cerebellar function. Adverse drug reactions are evaluated based on CTCAE version 4.0.

DETAILED DESCRIPTION:
1. Patients taking Nilotinib 1-1.Baseline information: demographics, genetic type of SCA, brain MRI, electrocardiography, routine blood evaluations 1-2. Time point of evaluation: At initiation of taking Nilotinib, 1, 3, 6, and 12 months 1-3. Evaluation items (at each time point) Routine check-up: electrocardiography, routine blood evaluations Adverse events: CTCAE version 4.0 Daily living performance: Barthel index General function: Friedreich's ataxia I and II 1-4. Change of drug dose Based on the attending physician's decision
2. Patients planning to take Nilotinib 2-1.Baseline information: demographics, genetic type of SCA, brain MRI, electrocardiography, routine blood evaluations 2-2. Time point of evaluation: Baseline, 1, 3, 6, and 12 months 2-3. Evaluation items (at each time point) Routine check-up: electrocardiography, routine blood evaluations Adverse events: CTCAE version 4.0 Cerebellar function: Scale for assessment and rating of ataxia (SARA) Daily living performance: Barthel index General function: Friedreich's ataxia I and II 2-4. Change of drug dose Based on the attending physician's decision

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as chronic cerebellar ataxia
* Confirmed as spinocerebellar ataxia by gene test

Exclusion Criteria:

* Laboratory abnormalities that could interfere with the proper use of Nilotinib QTc interval >450ms on initial electrocardiograph, Hb <8.0, WBC<2000, ANC <1600, PLT <140,000, AST >200, ALT>200, ALP>575, Positive HIV serology, active hepatitis B
* Unstable mental or physical status that could interfere with precise evaluation and proper management of SCA Heart failure (NYHA Grade III or IV), history of major heart disease Pregnancy, on breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Activity of daily living | 12 month
  Barthel index: score range 0-6

SECONDARY OUTCOMES:
Cerebellar function | 12 month
  Scale for the assessment and rating of ataxia (SARA): score range 0-36
General function | 12 month
  Rating scale for Friedreich's ataxia I: score range 0-6
Activity of daily living | 12 month
  Rating scale for Friedreich's ataxia II: score range 0-36

OTHER OUTCOMES:
Occurrence of adverse events | Baseline, 1 month, 3 month, 6 month, 12 month
  CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The IPD will be provided upon request from any qualified investigator.

REFERENCES:
- [Result] Lee WJ, Moon J, Kim TJ, Jun JS, Lee HS, Ryu YJ, Lee ST, Jung KH, Park KI, Jung KY, Kim M, Lee SK, Chu K. The c-Abl inhibitor, nilotinib, as a potential therapeutic agent for chronic cerebellar ataxia. J Neuroimmunol. 2017 Aug 15;309:82-87. doi: 10.1016/j.jneuroim.2017.05.015. Epub 2017 May 24. PMID 28601294
- [Derived] Lee WJ, Moon J, Jang Y, Shin YW, Son H, Shin S, Jeon D, Han D, Lee ST, Park KI, Jung KH, Lee SK, Chu K. Nilotinib treatment outcomes in autosomal dominant spinocerebellar ataxia over one year. Sci Rep. 2024 Jul 15;14(1):16303. doi: 10.1038/s41598-024-67072-z. PMID 39009709